CLINICAL TRIAL: NCT07125430
Title: Efficacy of Shock Wave Treatment to Reduce Pain and Improve Functionality in Patients With Knee Osteoarthritis: Randomized Clinical Trial.
Brief Title: Shock Wave Treatment in Patients With Knee Osteoarthritis
Acronym: SWKO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guadarrama Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Código H.U.P.H.: PI 119/25
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
Keywords: shock waves, knee osteoarthritis, rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): In the control group, a strengthening exercise program will be carried out for three weeks.
  Interventions: Other: strengthening exercise
- intervention group (Active Comparator): In the intervention group, in addition to the strengthening exercise program, 3 sessions of shock wave therapy (PiezoWave 2 Control Unit, classification 93/42/EEC class IIb) will be conducted, at a frequency of one session per week.
  The parameters for shock wave therapy will be: frequency 4-6 Hz, intensity 0.11-0.35 mJ/mm2, and number of pulses 2000 (applied to the femoral condyle and tibial plateau).
  Interventions: Other: strengthening exercise; Other: shock wave

INTERVENTIONS:
Other: strengthening exercise — a strengthening exercise program will be carried out for three weeks
Other: shock wave — 3 sessions of shock wave therapy, frequency of one session per week
  Arms: intervention group

SUMMARY:
Introduction: Knee osteoarthritis represents a significant health problem due to its impact on the functionality and quality of life of patients. Its treatment can be pharmacological, non-pharmacological, or surgical. Recently, the chondroprotective potential of shockwave therapy has been evidenced.

Objective: To determine whether shockwave treatment combined with knee strengthening exercises is superior to knee strengthening exercises alone in reducing pain and improving function in patients with knee osteoarthritis.

Method: A randomized controlled trial with allocation concealment is proposed. Patients with knee pain secondary to knee osteoarthritis will participate during their hospital admission. Two groups will be formed: both will follow an exercise program for three weeks, and the intervention group will add a weekly shockwave session during that same period.

The main variable will be pain intensity; other variables include stiffness, functional capacity, degree of satisfaction, and data related to the application of therapy (frequency, intensity, number of pulses, side effects). Clinical data will also be collected such as reason for admission, age, sex, comorbidities, degree of dependency, walking ability, analgesia, use of assistive devices, and progress during treatment.

Applicability: The results could lead to a change in clinical practice, serving as a basis for modifying treatment protocols for knee osteoarthritis in medium-stay hospitals. Furthermore, they would provide additional scientific evidence on the efficacy of shock wave therapy for this condition.

DETAILED DESCRIPTION:
The research team will recruit participants who meet inclusion criteria and do not present exclusion criteria during their admission to the functional recovery unit. A team member will inform and invite the subject to participate in the study. The Patient Information Sheet will be provided to them. Patients who decide to participate will need to sign the Informed Consent. At that moment, they will be scheduled to begin rehabilitation according to the protocol proposed for the study. Before starting treatment, patients will be randomized into treatment groups: shockwave treatment combined with knee strengthening exercises (intervention group) and treatment with knee strengthening exercises (control group).

The Data Collection Notebook will be completed, which has been prepared by the research team. In order to ensure the confidentiality of clinical data, these will be coded by dissociating the identifying and personal data from those necessary for the configuration of variables. For this, the principal investigator will carry out a coding process of the units of analysis.

All study participants will be evaluated at four points in time: before starting rehabilitative treatment, at the end of the three weeks of treatment, one month after the last treatment session, and three months after the last treatment session. At these four points, pain will be assessed using the VAS scale and functionality will be assessed using the WOMAC questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain assessed according to the VAS scale, with a score equal to or greater than 4 in the last 3 months.
* Osteoarthritis grade 2 or 3 in the Kellgren-Lawrence classification.
* Informed consent signature

Exclusion Criteria:

* Stroke in the last 3 months, knee surgery in the last 3 months, intra-articular infiltration in the last 3 months, secondary knee osteoarthritis, chronic inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Compare the magnitude of pain reduction between patients with knee osteoarthritis treated with shockwave therapy plus strengthening exercises and those treated only with strengthening exercises | From inclusion in the study until three months after the last treatment session
  To assess pain, the validated Visual Analog Scale (VAS) will be used. This scale represents pain intensity on a 10 cm horizontal line, where 0 corresponds to "no pain" and 10 to "the worst pain imaginable." The scores will be interpreted as follows: a score below 4 indicates mild or mild-to-moderate pain; a score between 4 and 6 suggests moderate to severe pain; and a score above 6 reflects the presence of intense or very severe pain.

SECONDARY OUTCOMES:
To examine difference in knee functionality improvement between both treatment groups | From inclusion in the study until three months after the last treatment session.
  To assess functionality, the Western Ontario and McMaster Universities Arthritis Index (WOMAC) questionnaire will be used. This instrument consists of 24 items grouped into three subscales: a pain subscale (5 items), a stiffness subscale (2 items), and a physical function subscale (17 items). Each item is rated using a 5-point Likert scale coded as follows: None = 0, Slight = 1, Moderate = 2, Severe = 3, and Extreme = 4. The scores for each subscale are summed separately, with a maximum of 20 points for pain, 8 for stiffness, and 68 for physical function. Higher scores indicate worse symptoms or greater disability, whereas lower scores reflect better condition or less impairment.
To evaluate the difference in degree of disability | From inclusion in the study until three months after the last treatment session.
  To evalute the difference in degree of disability between patients with knee osteoarthritis treated with shock wave therapy plus strengthening exercises and those treated with strengthening exercises alone. Lequesne Algofunctional Index will be used to assess the degree of functional disability associated with osteoarthritis. This validated questionnaire consists of 11 items distributed across three domains: pain or discomfort, maximum walking distance, and activities of daily living. The total score ranges from 0 to 24, with higher scores indicating greater severity of disability.
Analyze the level of patient satisfaction with the outcomes obtained from each therapeutic modality. | From inclusion in the study until three months after the last treatment session
  To evaluate the difference in degree of satisfaction (assessed using the Roles-Maudsley scale). Patient satisfaction will be assessed using the Roles and Maudsley scale, a four-point subjective rating system. Scores range from 1 (excellent) to 4 (poor), with lower scores indicating better outcomes. This scale reflects the patient's perception of pain relief and functional recovery after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yunia H Labrada Rodríguez, MD, MSc, Principal Investigator — Guadarrama Hospital
Locations (2):
- Spain (2):
  - Guadarrama Hospital, Guadarrama, Madrid
  - Hospital Guadarrama, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang CJ, Cheng JH, Chou WY, Hsu SL, Chen JH, Huang CY. Changes of articular cartilage and subchondral bone after extracorporeal shockwave therapy in osteoarthritis of the knee. Int J Med Sci. 2017 Feb 23;14(3):213-223. doi: 10.7150/ijms.17469. eCollection 2017. PMID 28367081
- [Background] Liao CD, Huang YY, Chen HC, Liou TH, Lin CL, Huang SW. Relative Effect of Extracorporeal Shockwave Therapy Alone or in Combination with Noninjective Treatments on Pain and Physical Function in Knee Osteoarthritis: A Network Meta-Analysis of Randomized Controlled Trials. Biomedicines. 2022 Jan 28;10(2):306. doi: 10.3390/biomedicines10020306. PMID 35203516
- [Background] Avendano-Coy J, Comino-Suarez N, Grande-Munoz J, Avendano-Lopez C, Gomez-Soriano J. Extracorporeal shockwave therapy improves pain and function in subjects with knee osteoarthritis: A systematic review and meta-analysis of randomized clinical trials. Int J Surg. 2020 Oct;82:64-75. doi: 10.1016/j.ijsu.2020.07.055. Epub 2020 Aug 13. PMID 32798759
- [Background] Wang CJ, Wang FS, Yang KD, Weng LH, Hsu CC, Huang CS, Yang LC. Shock wave therapy induces neovascularization at the tendon-bone junction. A study in rabbits. J Orthop Res. 2003 Nov;21(6):984-9. doi: 10.1016/S0736-0266(03)00104-9. PMID 14554209
- [Background] Chen YJ, Wang CJ, Yang KD, Kuo YR, Huang HC, Huang YT, Sun YC, Wang FS. Extracorporeal shock waves promote healing of collagenase-induced Achilles tendinitis and increase TGF-beta1 and IGF-I expression. J Orthop Res. 2004 Jul;22(4):854-61. doi: 10.1016/j.orthres.2003.10.013. PMID 15183445
- [Background] Berta L, Fazzari A, Ficco AM, Enrica PM, Catalano MG, Frairia R. Extracorporeal shock waves enhance normal fibroblast proliferation in vitro and activate mRNA expression for TGF-beta1 and for collagen types I and III. Acta Orthop. 2009 Oct;80(5):612-7. doi: 10.3109/17453670903316793. PMID 19916698
- [Background] Mittermayr R, Hartinger J, Antonic V, Meinl A, Pfeifer S, Stojadinovic A, Schaden W, Redl H. Extracorporeal shock wave therapy (ESWT) minimizes ischemic tissue necrosis irrespective of application time and promotes tissue revascularization by stimulating angiogenesis. Ann Surg. 2011 May;253(5):1024-32. doi: 10.1097/SLA.0b013e3182121d6e. PMID 21372687
- [Background] Uysal A, Yildizgoren MT, Guler H, Turhanoglu AD. Effects of radial extracorporeal shock wave therapy on clinical variables and isokinetic performance in patients with knee osteoarthritis: a prospective, randomized, single-blind and controlled trial. Int Orthop. 2020 Jul;44(7):1311-1319. doi: 10.1007/s00264-020-04541-w. Epub 2020 Mar 26. PMID 32215674
- [Background] ESWT Guidelines English version Updated and agreed from the ISMST Managing Board, in close cooperation with the Germanspeaking Society for Extracorporeal Shockwave Therapy (DIGEST) Daegu, South Korea July 20th, 2023 .ISMST-Guidelines-for-ESWT-_-engl-20240103.pdf
- [Background] Moya D, Ramon S, Schaden W, Wang CJ, Guiloff L, Cheng JH. The Role of Extracorporeal Shockwave Treatment in Musculoskeletal Disorders. J Bone Joint Surg Am. 2018 Feb 7;100(3):251-263. doi: 10.2106/JBJS.17.00661. No abstract available. PMID 29406349
- [Background] An S, Li J, Xie W, Yin N, Li Y, Hu Y. Extracorporeal shockwave treatment in knee osteoarthritis: therapeutic effects and possible mechanism. Biosci Rep. 2020 Nov 27;40(11):BSR20200926. doi: 10.1042/BSR20200926. PMID 33074309
- [Background] Giaretta S, Magni A, Migliore A, Natoli S, Puntillo F, Ronconi G, Santoiemma L, Sconza C, Viapiana O, Zanoli G. A Review of Current Approaches to Pain Management in Knee Osteoarthritis with a Focus on Italian Clinical Landscape. J Clin Med. 2024 Aug 31;13(17):5176. doi: 10.3390/jcm13175176. PMID 39274389
- [Background] Jhan SW, Wang CJ, Wu KT, Siu KK, Ko JY, Huang WC, Chou WY, Cheng JH. Comparison of Extracorporeal Shockwave Therapy with Non-Steroid Anti-Inflammatory Drugs and Intra-Articular Hyaluronic Acid Injection for Early Osteoarthritis of the Knees. Biomedicines. 2022 Jan 18;10(2):202. doi: 10.3390/biomedicines10020202. PMID 35203417